CLINICAL TRIAL: NCT03993392
Title: An Open-label, Rapid Initiation Study for Extended-Release Buprenorphine Subcutaneous Injection (SUBLOCADE)
Brief Title: SUBLOCADE Rapid Initiation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDV-6000-403
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine; Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TM buprenorphine followed by SUBLOCADE 300 mg (Experimental): Participants with a diagnosis of OUD stopped use of their current opioid prior to coming to the clinic to be assessed for withdrawal symptoms. If confirmed to be in withdrawal, participants were administered 4 mg transmucosal (TM) buprenorphine. If tolerated without sensitivity, clinical signs of sedation, or precipitated withdrawal, 300 mg SUBLOCADE was administered. Following SUBLOCADE administration, participants remained in the clinic for approximately 48 hours and were assessed for safety and tolerability, as well as for any signs of precipitated withdrawal. Participants returned to the clinic weekly, until the end-of-treatment (EOT) visit (28 days after SUBLOCADE administration).
  Interventions: Drug: TM buprenorphine; Drug: SUBLOCADE

INTERVENTIONS:
Drug: TM buprenorphine — 4mg TM buprenorphine, investigator choice as to brand
  Other Names: suboxone; subutex; belbuca; zubsolv; bunavail; generic buprenorphine
Drug: SUBLOCADE — 300mg subcutaneous injection
  Other Names: extended release buprenorphine

SUMMARY:
This study is to evaluate the safety and tolerability of initiating SUBLOCADE™ treatment following a shorter period of transmucosal (TM) buprenorphine treatment.

DETAILED DESCRIPTION:
Currently patients who are appropriate candidates for SUBLOCADE™ injection for subcutaneous (SC) use must initiate treatment with TM buprenorphine for a minimum of 7 days before receiving their first injection. This study is to evaluate the safety and tolerability of starting SUBLOCADE treatment following a shorter period.

Adults with moderate to severe opioid use disorder (OUD) not currently receiving medication assisted treatment will be recruited to participate. Prior to receiving TM buprenorphine, subjects will report their last opioid use and be experiencing at least mild withdrawal. Subjects will receive at least one dose of TM buprenorphine to ensure tolerability and that they show no evidence of precipitated withdrawal. If no evidence of intolerability or no precipitated withdrawal occurs, subjects will receive a single injection of SUBLOCADE and remain in the clinic for approximately 48 hours after the injection to assess for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF) and have the ability to comply with the requirements and restrictions listed therein.
* Documented history of moderate or severe opioid use disorder (OUD) as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
* Seeking buprenorphine-assisted treatment for OUD and is an appropriate candidate in the opinion of the Investigator or medically qualified sub-Investigator.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin test), is not lactating and, if of childbearing potential, agrees not to become pregnant while on the study and use medically acceptable means of contraception while on the study.

Exclusion Criteria:

* Current diagnosis, other than OUD, requiring chronic opioid treatment.
* Meet DSM-5 criteria for severe alcohol-use disorder.
* Has received any medication assisted treatment within 2 weeks.
* Concurrent or prior treatment with any long-acting depot form of buprenorphine containing products.
* Concurrent treatment with another investigational agent or enrolment in another clinical study (except for an observational study) or treatment with another investigational agent within 30 days prior to screening.
* Concurrent treatment with medications contraindicated for use with buprenorphine as per local prescribing information, including benzodiazepines or any other central nervous system depressants.
* Significant traumatic injury, major surgical procedure (as defined by the Investigator) within 30 days prior to Day 1 or still recovering from prior surgery.
* Any other active medical condition, organ disease or concurrent medication or treatment that may either compromise subject safety or interfere with study endpoints.
* Congenital long QT syndrome, history of prolonged QT in the 3 months prior to screening, or a corrected QT interval (Fridericia's - QTcF) >450 msec (male) or >470 msec (female), or history of risk factors for Torsades de Pointes. Known personal and/or family history of congenital QT prolongation, or taking Class IA antiarrhythmic medications (e.g., quinidine, procainamide, disopyramide) or Class III antiarrhythmic medications (e.g., sotalol, amiodarone) or other mediations that prolong the QT interval. Known family history of sudden unexplained death.
* Total bilirubin ≥1.5*upper limit of normal (ULN), alanine aminotransferase (ALT) ≥3*ULN, aspartate aminotransferase (AST) ≥5*ULN, serum creatinine >2*ULN at screening.
* Abdominal area unsuitable for SC injections.
* Uncontrolled intercurrent illness including, but not limited to, a medical or psychiatric illness/social situation that would limit compliance with study requirements or compromise the ability of the subject to provide written informed consent.
* Known allergy or hypersensitivity to buprenorphine, ATRIGEL or their excipients.
* Subject to court order requiring treatment for OUD.
* Subjects who are unable, in the opinion of the Investigator or Indivior, to comply fully with the study requirements including those who are currently incarcerated or pending incarceration/legal action.
* Clinic staff and/or subjects who have a financial interest in the study or who have an immediate family member of either the clinic staff and/or Indivior employees directly involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hassman, Principal Investigator — Hassman Research Institute
Locations (1):
- Hassman Research Institute, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hassman H, Strafford S, Shinde SN, Heath A, Boyett B, Dobbins RL. Open-label, rapid initiation pilot study for extended-release buprenorphine subcutaneous injection. Am J Drug Alcohol Abuse. 2023 Jan 2;49(1):43-52. doi: 10.1080/00952990.2022.2106574. Epub 2022 Aug 24. PMID 36001871
- [Result] Mariani JJ, Dobbins RL, Heath A, Gray F, Hassman H. Open-label investigation of rapid initiation of extended-release buprenorphine in patients using fentanyl and fentanyl analogs. Am J Addict. 2024 Jan;33(1):8-14. doi: 10.1111/ajad.13484. Epub 2023 Nov 8. PMID 37936553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 49 participants were screened and a total of 26 (53.1%) were enrolled into the study (i.e., were administered TM buprenorphine in the induction phase).
Pre-assignment Details: Reasons not enrolled:
  * 10 patients did not meet inclusion/exclusion criteria;
  * 3 did not meet Day 1 check-in criteria;
  * 3 withdrew consent;
  * 3 were not entered because the study was closed to enrolment;
  * 4 patients were for other reasons
Groups:
- TM Buprenorphine Followed by SUBLOCADE 300 mg: Participants with a diagnosis of opioid use disorder (OUD) stopped use of their current opioid prior to coming to the clinic to be assessed for withdrawal symptoms. If confirmed in withdrawal, participants were administered 4 mg transmucosal (TM) buprenorphine. If tolerated without sensitivity, clinical signs of sedation, or precipitated withdrawal, 300 mg SUBLOCADE was administered. Following SUBLOCADE administration, participants remained in the clinic for approximately 48 hours and were assessed for safety and tolerability, as well as for any signs of precipitated withdrawal. Participants returned to the clinic weekly, until the end-of-treatment (EOT) visit (28 days after SUBLOCADE administration).
Period: Overall Study
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Started | 26
Treated With SUBLOCADE (Safety and Full Analysis Sets) | 24
Completed | 20
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Did not meet Day 1 check-in criteria | 1

BASELINE CHARACTERISTICS:
Population: Safety and Full Analysis sets (same participants in each population)
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 9
  White | 13
  Other | 1
Age Group [Count of Participants; unit: Participants]
  >=18 to <30 years | 7
  >=30 to <45 years | 8
  >=45 to < 60 years | 6
  >=60 to < 65 years | 3
  >= 65 years | 0
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 22
  Not Reported | 2
Screening Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.60 (4.058)
Screening BMI Group [Count of Participants; unit: Participants] — Value ranges offered in units of kg/m^2.
  Participants
    0 to <18.5 (underweight) | 2
    >=18.5 and <25 (normal) | 18
    >=25 and <30 (overweight) | 1
    >=30 (obesity) | 3
Tobacco Use [Count of Participants; unit: Participants]
  Never | 2
  Current | 22
Caffeine Use [Count of Participants; unit: Participants]
  Never | 2
  Current | 22
Clinical Opiate Withdrawal Scale (COWS) Total Score at Screening [Mean (Standard Deviation); unit: units on a scale] — COWS is an 11-item instrument used to assess signs and symptoms of opioid withdrawal. The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderately severe withdrawal, and 37-48 severe withdrawal.
  units on a scale | 4.7 (4.63)
Opioid Craving Visual Analog Scale (OC-VAS) at Screening [Mean (Standard Deviation); unit: units on a scale] — The opioid craving scale was a 100 mm scale with 'no craving' indicated by 0 mm and 'strongest craving ever' indicated by 100 mm. Participants marked where along the scale reflected their craving for opioids.
  units on a scale | 58.3 (23.97)
Urine Drug Screen (UDS) for Opioids at Screening [Count of Participants; unit: Participants] — A participant was considered positive for opioids if the Screening Visit qualitative urine drug screen was positive for any of the substances: opioids, methadone, fentanyl, oxycodone or morphine.
  Participants
    Positive | 18
    Negative | 6
Opioid Drug Use History - Lifetime Use [Mean (Standard Deviation); unit: years] | 13.88 (13.542)
Opioid Drug Use History - Last 30 Days Use [Mean (Standard Deviation); unit: days] — Maximum number of days of use in last 30 days across all drugs within the class.
  days | 28.88 (3.837)
Opioid Drug Use History - Participants Use Intravenously in Last 30 Days [Count of Participants; unit: Participants] | 6
Day 1 Urine Drug Screen: Participants with Positive Opioid Tests [Count of Participants; unit: Participants]
  Morphine | 5
  Methadone | 1
  Fentanyl | 17
  Oxycodone | 3

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Experienced Any Precipitated Withdrawal Within One Hour After SUBLOCADE Administration
Description: Clinical Opiate Withdrawal Scale (COWS) is an 11-item instrument used to assess signs and symptoms of opioid withdrawal. The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderately severe withdrawal, and 37-48 severe withdrawal.
  Precipitated withdrawal was defined as in increase in Clinical Opioid Withdrawal Scale (COWS) score by ≥6 from the pre-SUBLOCADE value within 1 hour SUBLOCADE injection.
Time Frame: Day 1: Pre-SUBLOCADE evaluation taken after TM buprenorphine treatment and prior to injection: SUBLOCADE evaluation taken within one hour of SUBLOCADE injection
Population: Full analysis set (FAS): Participants who receive a SUBLOCADE injection and have data for >=1 COWS assessment at the Pre-SUBLOCADE timepoint just before the SUBLOCADE injection and a COWS assessment within one hour after the SUBLOCADE injection. One participant did not have a COWS score at one hour so is not included.
Measure: Count of Participants; unit: Participants
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 23
Participants | 1

2. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: A TEAE was an AE that started after the administration of TM buprenorphine for induction on Day 1.
  TEAE=any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator as mild, moderate and severe, with severe= a marked limitation in activity. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical or surgical intervention to prevent one of the outcomes listed in this definition. AEs of special interest include SUBOCADE depot removal, occurrences of alanine aminotransferase (ALT) >3*upper limit of normal (ULN) and bilirubin >2*ULN.
Time Frame: Day 1 to Day 28
Population: The safety population was used for the safety analysis, and consisted of all participants who received at least 1 dose of SUBLOCADE
Measure: Count of Participants; unit: Participants
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 24
Participants
  Any TEAE | 20
  Study Drug-related TEAE | 5
  Serious TEAE | 0
  Related and Serious TEAE | 0
  Severe TEAE | 5
  TEAE leading to death | 0
  TEAE leading to discontinuation of drug | 0
  TEAE leading to interruption of drug | 0
  Serious TEAEs - discontinuation of drug | 0
  Serious TEAEs - interruption of drug | 0
  AE of Special Interest | 0

3. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE) Within 48 Hours Post-SUBLOCADE Injection
Description: as for outcome 2
Time Frame: Day 1 SUBLOCADE injection up to 48 hours later
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 24
Participants
  Any TEAE | 19
  Study Drug-related TEAE | 4
  Serious TEAE | 0
  Related and Serious TEAE | 0
  Severe TEAE | 5
  TEAE leading to death | 0
  TEAE leading to discontinuation of drug | 0
  TEAE leading to interruption of drug | 0
  Serious TEAEs - discontinuation of drug | 0
  Serious TEAEs - interruption of drug | 0
  AE of Special Interest | 0

4. Secondary Outcome: Cumulative Number of Participants Who Experienced a >=6 Point Clinical Opiate Withdrawal Scale (COWS) Total Score Increase After SUBLOCADE Administration From the Pre-SUBLOCADE Value at Key Timepoints
Description: COWS is an 11-item instrument used to assess signs and symptoms of opioid withdrawal. The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderately severe withdrawal, and 37-48 severe withdrawal.
  Cumulative number of participants in key timepoints who had a COWS total score increase of ≥6 points from the pre-SUBLOCADE value.
Time Frame: Day 1: Pre-SUBLOCADE evaluation taken after TM buprenorphine treatment and prior to injection: SUBLOCADE evaluations taken 1, 6, 12, 24 and 48 hours after SUBLOCADE injection.
Population: Full analysis set (FAS) of participants 'at risk' at the start of the time interval. A participant was at risk if they had a pre-SUBLOCADE COWs assessment and COWS assessments at the current and all prior key timepoints and did not have the event in a previous timepoint. One participant did not have a COWS score at one hour so is not included.
Measure: Count of Participants; unit: Participants
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 23
Participants
  >0 to 1 hour | 1
  > 1 to 6 hours: number analyzed (Participants) | 21
  > 1 to 6 hours | 2
  >6 to 12 hours: number analyzed (Participants) | 13
  >6 to 12 hours | 2
  >12 to 24 hours: number analyzed (Participants) | 13
  >12 to 24 hours | 2
  >24 to 48 hours: number analyzed (Participants) | 13
  >24 to 48 hours | 2

5. Secondary Outcome: COWS Total Score Normalized Area Under the Curve (AUC) Through Key Timepoints Post SUBLOCADE Injection
Description: The area under the curve (AUC) for COWS total score from the pre-SUBLOCADE value to a later time point were calculated using the linear trapezoidal method. For each analysis time interval (AUC0-1hr, AUC0-6hrs, AUC0-12hrs, AUC0-24hrs, AUC0-48hrs) the AUC value was normalized across participants for the actual duration (in hours) of the time interval. The normalized AUC for COWS can be interpreted as the averaged AUC per hour or the averaged COWS over a time interval, as if the COWS was measured hourly during that time interval.
  Participants were included in a given interval if they had a pre-SUBLOCADE COWS assessment and a COWS assessment at the terminal timepoint for the interval.
Time Frame: SUBLOCADE injection on Day 1 through 1, 6, 12, 24 and 48 hours after SUBLOCADE injection
Population: Full analysis set. Participants were included in a given interval if they had a pre-SUBLOCADE COWS assessment and a COWS assessment at the terminal timepoint for the interval.
Measure: Mean (Standard Deviation); unit: hours*units on a scale
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 24
hours*units on a scale
  Through 1 hour post SUBLOCADE | 11.91 (3.700)
  Through 6 hours post SUBLOCADE: number analyzed (Participants) | 23
  Through 6 hours post SUBLOCADE | 9.27 (3.939)
  Through 12 hours post SUBLOCADE: number analyzed (Participants) | 23
  Through 12 hours post SUBLOCADE | 7.91 (3.772)
  Through 24 hours post SUBLOCADE: number analyzed (Participants) | 23
  Through 24 hours post SUBLOCADE | 6.59 (3.021)
  Through 48 hours post SUBLOCADE: number analyzed (Participants) | 23
  Through 48 hours post SUBLOCADE | 5.03 (2.566)

6. Secondary Outcome: Total Score on COWS At Timepoints During the Treatment Period
Description: Clinical Opiate Withdrawal Scale (COWS) is an 11-item instrument used to assess signs and symptoms of opioid withdrawal. The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderately severe withdrawal, and 37-48 severe withdrawal.
Time Frame: Day 1 to Day 29
Population: Full analysis set of participants with data at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 24
units on a scale
  Day 1 Check-in | 12.5 (3.74)
  Pre TM Buprenephrine | 14.6 (4.13)
  Pre-SUBLOCADE | 12.6 (4.05)
  1 hour post-SUBLOCADE dose: number analyzed (Participants) | 23
  1 hour post-SUBLOCADE dose | 11.1 (4.51)
  2 hours post-SUBLOCADE dose: number analyzed (Participants) | 22
  2 hours post-SUBLOCADE dose | 10.1 (4.99)
  3 hours post-SUBLOCADE dose: number analyzed (Participants) | 19
  3 hours post-SUBLOCADE dose | 9.1 (5.32)
  4 hours post-SUBLOCADE dose: number analyzed (Participants) | 21
  4 hours post-SUBLOCADE dose | 8.0 (3.93)
  6 hours post-SUBLOCADE dose: number analyzed (Participants) | 22
  6 hours post-SUBLOCADE dose | 6.9 (4.06)
  8 hours post-SUBLOCADE dose: number analyzed (Participants) | 19
  8 hours post-SUBLOCADE dose | 6.6 (3.83)
  12 hours post-SUBLOCADE dose: number analyzed (Participants) | 16
  12 hours post-SUBLOCADE dose | 6.6 (3.69)
  16 hours post-SUBLOCADE dose: number analyzed (Participants) | 3
  16 hours post-SUBLOCADE dose | 6.0 (2.65)
  20 hours post-SUBLOCADE dose: number analyzed (Participants) | 16
  20 hours post-SUBLOCADE dose | 5.0 (2.90)
  24 hours post-SUBLOCADE dose: number analyzed (Participants) | 22
  24 hours post-SUBLOCADE dose | 4.2 (3.16)
  30 hours post-SUBLOCADE dose: number analyzed (Participants) | 20
  30 hours post-SUBLOCADE dose | 3.9 (3.00)
  36 hours post-SUBLOCADE dose: number analyzed (Participants) | 19
  36 hours post-SUBLOCADE dose | 3.5 (2.65)
  48 hours post-SUBLOCADE dose: number analyzed (Participants) | 23
  48 hours post-SUBLOCADE dose | 2.8 (2.54)
  Day 8: number analyzed (Participants) | 22
  Day 8 | 1.9 (1.64)
  Day 15: number analyzed (Participants) | 22
  Day 15 | 2.0 (1.99)
  Day 22: number analyzed (Participants) | 20
  Day 22 | 2.0 (2.58)
  End of Treatment Day 29: number analyzed (Participants) | 21
  End of Treatment Day 29 | 1.8 (2.12)

7. Secondary Outcome: Total Score on Opioid Craving Visual Analogue Scale (OC-VAS) At Timepoints During the Treatment Period
Description: Participants indicated their level of craving for opioids by marking a 100mm visual analogue scale where 0 = no craving and 100 = maximal craving.
Time Frame: Day 1 to Day 29
Population: Full analysis set of participants with data at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TM Buprenorphine Followed by SUBLOCADE 300 mg
Number analyzed (Participants) | 24
units on a scale
  Day 1 Check-in | 66.0 (22.03)
  Pre TM Buprenephrine | 65.0 (31.06)
  Pre-SUBLOCADE | 57.0 (28.91)
  1 hour post-SUBLOCADE dose: number analyzed (Participants) | 22
  1 hour post-SUBLOCADE dose | 56.5 (26.52)
  2 hours post-SUBLOCADE dose: number analyzed (Participants) | 22
  2 hours post-SUBLOCADE dose | 52.8 (29.99)
  3 hours post-SUBLOCADE dose: number analyzed (Participants) | 19
  3 hours post-SUBLOCADE dose | 53.9 (30.22)
  4 hours post-SUBLOCADE dose: number analyzed (Participants) | 21
  4 hours post-SUBLOCADE dose | 44.5 (29.75)
  6 hours post-SUBLOCADE dose: number analyzed (Participants) | 22
  6 hours post-SUBLOCADE dose | 42.6 (26.98)
  8 hours post-SUBLOCADE dose: number analyzed (Participants) | 19
  8 hours post-SUBLOCADE dose | 43.1 (27.20)
  12 hours post-SUBLOCADE dose: number analyzed (Participants) | 16
  12 hours post-SUBLOCADE dose | 39.3 (31.19)
  16 hours post-SUBLOCADE dose: number analyzed (Participants) | 3
  16 hours post-SUBLOCADE dose | 29.7 (38.48)
  20 hours post-SUBLOCADE dose: number analyzed (Participants) | 16
  20 hours post-SUBLOCADE dose | 33.5 (20.79)
  24 hours post-SUBLOCADE dose: number analyzed (Participants) | 22
  24 hours post-SUBLOCADE dose | 27.3 (20.77)
  30 hours post-SUBLOCADE dose: number analyzed (Participants) | 20
  30 hours post-SUBLOCADE dose | 16.7 (12.37)
  36 hours post-SUBLOCADE dose: number analyzed (Participants) | 19
  36 hours post-SUBLOCADE dose | 13.8 (13.74)
  48 hours post-SUBLOCADE dose: number analyzed (Participants) | 23
  48 hours post-SUBLOCADE dose | 12.1 (12.09)
  Day 8: number analyzed (Participants) | 22
  Day 8 | 7.6 (11.00)
  Day 15: number analyzed (Participants) | 22
  Day 15 | 6.4 (9.54)
  Day 22: number analyzed (Participants) | 20
  Day 22 | 13.1 (20.32)
  End of Treatment Day 29: number analyzed (Participants) | 21
  End of Treatment Day 29 | 7.3 (9.24)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 29
Groups:
- Induction Phase: Treatment-emergent adverse events (TEAEs) where the start date/time of the event is on or after the date/time of the administration of transmucosal (TM) buprenorphine (BUP) for induction but prior to the date/time of the SUBLOCADE injection.
- Safety Population (Post -SUBLOCADE): Treatment-emergent adverse events (TEAEs) where the start date/time of the event is post-SUBLOCADE injection.
Arm/Group | Induction Phase | Safety Population (Post -SUBLOCADE)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 4/26 | 20/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase (N=26) | Safety Population (Post -SUBLOCADE) (N=24)
Irritability (Psychiatric disorders) | 0 | 12
Anxiety (Psychiatric disorders) | 2 | 9
Insomnia (Psychiatric disorders) | 0 | 6
Agitation (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 10
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 1 | 3
Pain (General disorders) | 2 | 8
Chills (General disorders) | 0 | 3
Injection site bruising (General disorders) | 0 | 3
Injection site erythema (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infusion site cellulitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multicenter publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.

DOCUMENTS (2):
  • Study Protocol (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03993392/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03993392/SAP_001.pdf